CLINICAL TRIAL: NCT00799877
Title: A 10-Year, Post-marketing, Observational Study to Assess Long Term Safety of HUMIRA® (Adalimumab) in Adult Patients With Chronic Plaque Psoriasis (PS)
Brief Title: Chronic Plaque Psoriasis (Ps) Registry
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P10-023
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Psoriasis; Moderate Psoriasis; Severe Psoriasis; Chronic Plaque Psoriasis; Severe Chronic Plaque Psoriasis; Registry
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1: This registry will evaluate the long-term safety and effectiveness of HUMIRA® as used in routine clinical practice.

SUMMARY:
The purpose of this study is to evaluate the long-term safety of Humira® in Adult Patients with Chronic Plaque Psoriasis (Ps).

DETAILED DESCRIPTION:
ESPRIT is a 10 year registry of patients taking HUMIRA® for Psoriasis. Patients who volunteer to participate will be asked to provide information about their medical history and experiences with HUMIRA®. No registry specific testing will be performed. Patients will be asked to provide data on their experiences with HUMIRA® approximately every 6 months, or as determined by the study doctor. No drug will be provided as a result of participation in the registry. All treatment decisions are independent of participation in the registry.

ELIGIBILITY:
Inclusion Criteria:

1. An adult patient (18 years of age or older) with chronic plaque psoriasis who has been prescribed HUMIRA® therapy according to the local product labeling and meets one of the following criteria:

   * New initiated (within 4 weeks of registry entry) on HUMIRA® therapy;
   * Initiated HUMIRA® therapy in the past and:

     * Has received continuous (no more than 70 consecutive days off drug) HUMIRA® therapy and the physician can provide source documentation of SAEs, AEs, of Special Interest, and dosing information since initiation of therapy.

   OR
   * Is entering after participation in an AbbVie HUMIRA (adalimumab) sponsored study and has received continuous (no more than 70 consecutive days off drug) HUMIRA® therapy after the completion of AbbVie sponsored study and physician can provide source documentation of SAEs, AEs of Special Interest, and dosing information since initiation of commercial HUMIRA® (defined as a prescribed/non study drug).
2. Patient is willing to consent to data being collected and provided to AbbVie;
3. Patient is capable of and willing to give written informed consent and to comply with the requirements of the registry.

Exclusion Criteria:

- Patient should not be enrolled if he/she cannot be treated in accordance with the local product label.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, departments of dermatology
Sampling Method: Non-Probability Sample
Enrollment: 6065 (Actual)
Dates: Start 2008-09-26 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events | Duration of study
  Incidence of Adverse Events is calculated upon all events that occur during registry, during exposure to HUMIRA® prior to entry of registry, and in Health Care Provider process.
Incidence of Adverse Events of Special Interest | Duration of study
  Incidence of Adverse Events is calculated upon all events that occur during registry, during exposure to HUMIRA® prior to entry of registry, and in Health Care Provider process.
Adverse Events that lead to permanent discontinuation of HUMIRA® | Duration of study
  Incidence of Adverse Events that lead to permanent discontinuation of HUMIRA® is calculated upon all events that lead to permanent discontinuation of HUMIRA® during registry, during exposure to HUMIRA® prior to entry of registry, and in Health Care Provider process.

SECONDARY OUTCOMES:
Health Care Utilization | Duration of study
Work Productivity and Activity Impairment Questionnaire: Specific Health Problem | Duration of study
Patient Global Assessment | Duration of study
Patient Health Question-9 | Duration of study
Medical Outcomes Social Activities Scale | Duration of study
Patient reported outcome - Dermatology Life Quality Index | Duration of study
Census | Duration of study
Psoriasis Impact and Experience | Duration of study
Illness Cognition | Duration of study
Insurance Status | Duration of study
Rosenberg Self-Esteem Scale | Duration of study
Physician's Global Assessment | Collected approximately every six months.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (339):
- United States (222):
  - Southview Medical Group, PC /ID# 20961, Birmingham, Alabama
  - Total Skin and Beauty Derm Ctr /ID# 17156, Birmingham, Alabama
  - Inverness Dermatology /ID# 76194, Birmingham, Alabama
  - McLain Medical Associates, PC /ID# 18351, Birmingham, Alabama
  - Deep South Dermatology, PC /ID# 40267, Daphne, Alabama
  - Northeast Alabama Dermatology /ID# 76193, Huntsville, Alabama
  - Yates, Huntsville, AL /ID# 17130, Huntsville, Alabama
  - Mobile Dermatology, P.C. /ID# 19783, Mobile, Alabama
  - Medical Dermatology Specialist /ID# 76113, Phoenix, Arizona
  - Arizona Advanced Dermatology /ID# 20512, Phoenix, Arizona
  - Camelback Dermatology & Skin Surgery /ID# 18901, Phoenix, Arizona
  - Alliance Dermatology and MOHs Center, PC /ID# 17087, Phoenix, Arizona
  - Omni Dermatology Research /ID# 135562, Phoenix, Arizona
  - Affiliated Dermatology /ID# 18327, Scottsdale, Arizona
  - Specialists in Dermatology /ID# 18864, Tucson, Arizona
  - Johnson Dermatology Clinic /ID# 17088, Fort Smith, Arkansas
  - Hull Dermatology, PA /ID# 17086, Rogers, Arkansas
  - Elite MD Adv Derm Laser /ID# 28323, Danville, California
  - Center for Dermatology Clinical Research /ID# 20722, Fremont, California
  - Associates in Research /ID# 17544, Fresno, California
  - Dermatology and Dermatologic /ID# 17145, Garden Grove, California
  - Guagenti, Glendale, CA /ID# 28263, Glendale, California
  - Miremadi Dermatology /ID# 24323, La Jolla, California
  - SCRIPPS Clinic /ID# 28147, La Mesa, California
  - Dr. Abdallah Khourdaji /ID# 24307, Lodi, California
  - Premiere Clinical Research,LLC /ID# 44719, Long Beach, California
  - Kaiser Permanente LA Med Ctr /ID# 24334, Los Angeles, California
  - Dermatology Research Associates /ID# 17158, Los Angeles, California
  - California Skin Institute /ID# 19769, Mountain View, California
  - Quest Dermatology Research /ID# 71677, Northridge, California
  - Dermatology Medical Group of Oxnard /ID# 17102, Oxnard, California
  - Univ California, San Francisco /ID# 28267, San Francisco, California
  - Danesh, San Gabriel, CA /ID# 23068, San Gabriel, California
  - Carson, San Jose, CA /ID# 17064, San Jose, California
  - East Bay Psoriasis Trmnt Ctr /ID# 17081, San Ramon, California
  - Redwood Family Dermatology /ID# 76119, Santa Rosa, California
  - Skin Physicians & Surgeons Med /ID# 40265, Upland, California
  - Advanced Dermatology & Cosmetic Care /ID# 20511, Valencia, California
  - Solano Dermatology Associates /ID# 20727, Vallejo, California
  - Colorado Springs Derm Clinic /ID# 28165, Colorado Springs, Colorado
  - Skin Care Specialists of CO /ID# 17142, Longmont, Colorado
  - Moss and Maiocco, MD, LLC /ID# 69767, Bridgeport, Connecticut
  - Notaro, Danbury, CT /ID# 40264, Danbury, Connecticut
  - Derm Assoc of Western CT /ID# 71673, Danbury, Connecticut
  - Choi, New Haven, CT /ID# 58982, New Haven, Connecticut
  - Panzer Dermatology & Cosmetic /ID# 17131, Newark, Delaware
  - Panzer Dermatology & Cosmetic /ID# 17146, Newark, Delaware
  - George Washington University Hospital /ID# 24270, Washington D.C., District of Columbia
  - Private Practice- Dr. Tory Sullivan /ID# 17126, Aventura, Florida
  - Dermatology and Skin Surgery /ID# 88353, Celebration, Florida
  - Florida Academic Centers Research and Education /ID# 24273, Coral Gables, Florida
  - Dermatology Associates of the Palm Beaches /ID# 17137, Delray Beach, Florida
  - Ft. Lauderdale Derm & Cosmetic /ID# 23071, Fort Lauderdale, Florida
  - Hollywood Dermatology /ID# 17129, Hollywood, Florida
  - Hollywood Dermatology /ID# 19771, Hollywood, Florida
  - Suncoast Dermatology and Skin Surgery Center /ID# 23067, Lecanto, Florida
  - Athenea Assoc Med Research /ID# 69768, Miami, Florida
  - Assoc. in Med & Surg Derm /ID# 17523, Naples, Florida
  - Central Florida Dermatology Associates /ID# 20508, Orlando, Florida
  - Gulf Coast Dermatology /ID# 20724, Panama City, Florida
  - Snyder, Pembroke Pines, FL /ID# 17122, Pembroke Pines, Florida
  - Gary L. Heller - Dermatology Research Cosmetic Center /ID# 17083, Pinellas Park, Florida
  - Skin and Cancer Associates /ID# 20726, Plantation, Florida
  - The Center for Skin Wellness /ID# 42005, Sarasota, Florida
  - Water's Edge Dermatology - Stuart /ID# 76114, Stuart, Florida
  - Scannon, Tampa, Florida /ID# 28160, Tampa, Florida
  - University of South Florida /ID# 38289, Tampa, Florida
  - Ctr for Derm & Skin Surgery /ID# 28210, Tampa, Florida
  - Geisinger Medical Center /ID# 17521, Tampa, Florida
  - Coast Derm & Skin Cancer Ctr /ID# 40189, Venice, Florida
  - Heskel, Vero Beach, FL /ID# 69764, Vero Beach, Florida
  - Hamilton Research, LLC /ID# 20503, Alpharetta, Georgia
  - Parker, Atlanta, GA /ID# 40190, Atlanta, Georgia
  - Skin Cancer & Cosmetic Derm Ct /ID# 23313, Calhoun, Georgia
  - East Metro Dermatology PC /ID# 20505, Conyers, Georgia
  - Dermatologic Surgery Specialis /ID# 17149, Macon, Georgia
  - NW GA Dermatology & Skin Cancer Specialists /ID# 17089, Marietta, Georgia
  - Paula Nelson MD & Associates /ID# 23076, Marietta, Georgia
  - RI Dermatology & Cosmetic Ctr /ID# 40270, Newport, Georgia
  - Skin Cancer & Cosmetic Derm /ID# 24305, Rome, Georgia
  - Northwest Georgia Dermatology /ID# 28162, Rome, Georgia
  - Atlanta Derm & Laser Surgery /ID# 28144, Tucker, Georgia
  - Wray, Blackfoot, ID /ID# 24333, Blackfoot, Idaho
  - Idaho Skin Institute /ID# 76118, Chubbuck, Idaho
  - Saltzer Medical Group /ID# 17144, Nampa, Idaho
  - Olmstead, Twin Falls, ID /ID# 24325, Twin Falls, Idaho
  - Pinski Dermatology /ID# 17147, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine /ID# 28169, Chicago, Illinois
  - John H. Stroger, Jr. Hosp /ID# 40185, Chicago, Illinois
  - Rush University Medical Center /ID# 47604, Chicago, Illinois
  - Del Campo, Chicago, IL /ID# 19770, Chicago, Illinois
  - Lakeside Dermatology /ID# 247839, Libertyville, Illinois
  - Loyola University Medical Ctr /ID# 23065, Maywood, Illinois
  - Arlington Dermatology /ID# 23062, Rolling Meadows, Illinois
  - Schaumburg Dermatology, SC /ID# 38294, Schaumburg, Illinois
  - DuPage Medical Group /ID# 18861, Wheaton, Illinois
  - DuPage Medical Group /ID# 20507, Wheaton, Illinois
  - Mercy Woodstock Medical Center /ID# 40186, Woodstock, Illinois
  - Shideler Dermatology Group /ID# 69957, Carmel, Indiana
  - Spencer Dermatology Associates /ID# 71678, Crawfordsville, Indiana
  - Indiana University /ID# 37052, Indianapolis, Indiana
  - Dawes Fretzin, LLC /ID# 17151, Indianapolis, Indiana
  - Dawes Fretzin, LLC /ID# 17502, Indianapolis, Indiana
  - Dermatology Associates of Indiana /ID# 24269, Indianapolis, Indiana
  - The Dermatology Center PSC - New Albany /ID# 20501, New Albany, Indiana
  - The Indiana Clinical Trials Center /ID# 17153, Plainfield, Indiana
  - Great Plains Dermatology, P.A. /ID# 23079, Hays, Kansas
  - Epiphany Dermatology of Kansas LLC /ID# 19764, Overland Park, Kansas
  - Kansas Medical Clinic /ID# 28212, Topeka, Kansas
  - Knuckles, Corbin, KY /ID# 17101, Corbin, Kentucky
  - Anapolis Dermatology Center /ID# 24302, Annapolis, Maryland
  - Glassman, Bethesda, MD /ID# 17069, Bethesda, Maryland
  - Dermatology and Skin Cancer Specialists, LLC /ID# 65884, Rockville, Maryland
  - Charles County Dermatology /ID# 18341, White Plains, Maryland
  - Brigham Dermatology Associates /ID# 28207, Boston, Massachusetts
  - Worcester Dermatology Assoc. /ID# 37048, Worcester, Massachusetts
  - David Fivenson, MD, PLC /ID# 20504, Ann Arbor, Michigan
  - Iacobelli, Clinton Twnshp, MI /ID# 38290, Clinton Township, Michigan
  - Hamzavi Dermatology /ID# 25903, Fort Gratiot, Michigan
  - Pinnacle Dermatology - Grand Blanc /ID# 40196, Grand Blanc, Michigan
  - Stawiski, Grand Rapids, MI /ID# 17124, Grand Rapids, Michigan
  - Lakeshore Dermatology /ID# 24330, Norton Shores, Michigan
  - Somerset Skin Centre /ID# 17157, Troy, Michigan
  - St. Louis University /ID# 28150, St Louis, Missouri
  - Metro Hypertension and Kidney /ID# 40184, St Louis, Missouri
  - Dermatology Associates, Inc. /ID# 23075, St Louis, Missouri
  - Town Center Dermatology /ID# 28152, Wildwood, Missouri
  - Assoc. Derm & Skin Cancer Clin /ID# 24303, Helena, Montana
  - Center of Dermatology, P.C. /ID# 23078, Omaha, Nebraska
  - Academic Dermatology of Nevada /ID# 20513, Henderson, Nevada
  - Linda Woodson Dermatology /ID# 18333, Las Vegas, Nevada
  - Nathan Adelson Hospice /ID# 18332, Las Vegas, Nevada
  - Riley, Reno, NV /ID# 36343, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center /ID# 20502, Lebanon, New Hampshire
  - Nashua Dermatology /ID# 18352, Nashua, New Hampshire
  - Belleville Dermatology Center /ID# 17067, Belleville, New Jersey
  - Psoriasis Treatment Center of Central New Jersey /ID# 17148, East Windsor, New Jersey
  - Fernandez-Obregon, Hoboken, NJ /ID# 23073, Hoboken, New Jersey
  - Fulk, Morristown, TN /ID# 18344, Morristown, New Jersey
  - UMDNJ R. W. Johnson Med School /ID# 24326, Somerset, New Jersey
  - Derm Consultants of Summit /ID# 24308, Summit, New Jersey
  - The Dermatology Group, PC /ID# 28158, Verona, New Jersey
  - Marcus, Wyckoff, NJ /ID# 23074, Wyckoff, New Jersey
  - Reflections Dermatology & Psoriasis canter /ID# 19781, Auburn, New York
  - The Dermatology Center, PSC - Bayside NY /ID# 28170, Bayside, New York
  - Garden City Dermatology /ID# 42003, Garden City, New York
  - Bruckstein, Lawrence, NY /ID# 17063, Lawrence, New York
  - Scheinfeld, New York, NY /ID# 17136, New York, New York
  - New York Presbyterian Hospital Weill Cornell Medical Center /ID# 24268, New York, New York
  - South Nassau Dermatology /ID# 17065, Oceanside, New York
  - The Ctr for Derm at Lifetime /ID# 47603, Rochester, New York
  - Dermedx Dermatology, PC /ID# 28163, Smithtown, New York
  - Central Dermatology Center, PA /ID# 17070, Chapel Hill, North Carolina
  - Dr. Aida Lugo-Somolinos /ID# 24309, Chapel Hill, North Carolina
  - Fraser, Charlotte, NC /ID# 19772, Charlotte, North Carolina
  - Duke Cancer Center /ID# 24324, Durham, North Carolina
  - Piedmont Dermatology Center /ID# 18326, Greensboro, North Carolina
  - Dermatology Associates of Coastal Carolina /ID# 76116, New Bern, North Carolina
  - Carolina Skin Care /ID# 19773, Pinehurst, North Carolina
  - Andrus and Assoc Dermatology /ID# 20510, Raleigh, North Carolina
  - Boice-Willis Clinic, P.A. /ID# 17125, Rocky Mount, North Carolina
  - Crane, Wilmington, NC /ID# 17066, Wilmington, North Carolina
  - Wilmington Dermatology Center /ID# 69763, Wilmington, North Carolina
  - Polley Clinic of Dermatology /ID# 18334, Wilson, North Carolina
  - PMG Research of Winston-Salem /ID# 17133, Winston-Salem, North Carolina
  - Hawkins, Akron, Ohio /ID# 28149, Akron, Ohio
  - Summa Physicians Dermatology /ID# 37051, Akron, Ohio
  - Oakview Dermatology, LLC /ID# 38298, Athens, Ohio
  - Austintown /ID# 76121, Austintown, Ohio
  - The Ohio State University /ID# 43150, Columbus, Ohio
  - Allied Dermatology and Skin Surgery /ID# 28154, Fairlawn, Ohio
  - Brodell Medical Inc. /ID# 24304, Warren, Ohio
  - Univ Oklahoma HSC /ID# 28145, Oklahoma City, Oklahoma
  - Tulsa Dermatology Clinic, Inc. /ID# 71675, Tulsa, Oklahoma
  - Oregon Dermatology and Research Center /ID# 24327, Portland, Oregon
  - Oregon Medical Research Center /ID# 28143, Portland, Oregon
  - Altoona Ctr Clinical Res /ID# 17155, Duncansville, Pennsylvania
  - University of Pittsburgh MC /ID# 17068, Pittsburgh, Pennsylvania
  - Mikell, Beaufort, SC /ID# 17143, Beaufort, South Carolina
  - Hampton, Charleston, NC /ID# 18865, Charleston, South Carolina
  - Coastal Clinical Research Center of the Carolinas /ID# 18353, Charleston, South Carolina
  - Westside Dermatology, LLC /ID# 17541, Spartanburg, South Carolina
  - MidSouth Dermatology /ID# 17128, Bartlett, Tennessee
  - Skin Cancer & Cosmetic Derm /ID# 65882, Cleveland, Tennessee
  - Dermatology Associates /ID# 42008, Kingsport, Tennessee
  - Arlington Research Center, Inc /ID# 23063, Arlington, Texas
  - Austin Dermatology Associates /ID# 38296, Austin, Texas
  - Steiner Ranch Dermatology /ID# 20509, Austin, Texas
  - Dermatology Treatment and Research Center /ID# 17545, Dallas, Texas
  - Aftergut, Dallas, TX /ID# 17041, Dallas, Texas
  - Texas Dermatology Associates /ID# 28155, Dallas, Texas
  - Texas Dermatology Associates /ID# 28157, Dallas, Texas
  - Schwartz,Harlingen,TX,US /ID# 20725, Harlingen, Texas
  - Sonabend, Houston, TX /ID# 17123, Houston, Texas
  - Heights Dermatology & Aesthetic Center /ID# 28325, Houston, Texas
  - Memorial Clinical Associates /ID# 17085, Houston, Texas
  - West Houston Dermatology /ID# 18330, Houston, Texas
  - Lehman Dermatology Clinic /ID# 17082, Lubbock, Texas
  - Texas Tech University Health Sciences Center - Lubbock /ID# 37050, Lubbock, Texas
  - The Dermatology Inst of S. TX /ID# 38288, McAllen, Texas
  - Dermatology Associates of San Antonio /ID# 17150, San Antonio, Texas
  - Tucker, The Woodlands, Texas /ID# 38295, The Woodlands, Texas
  - Aspen Dermatology, PLLC /ID# 38293, Spanish Fork, Utah
  - Aspen Dermatology, PLLC /ID# 40183, Spanish Fork, Utah
  - Aspen Dermatology, PLLC /ID# 40192, Spanish Fork, Utah
  - Premier Dermatology /ID# 69958, Ashburn, Virginia
  - Skin and Laser Surgery Center /ID# 40182, Tysons Corner, Virginia
  - Tidewater Skin Care/Pathology /ID# 71674, Virginia Beach, Virginia
  - Dermatology & Laser Center NW /ID# 18324, Bellingham, Washington
  - Dermatology Associates of Seattle /ID# 18328, Seattle, Washington
  - Dermatology Associates of Seattle /ID# 19802, Seattle, Washington
  - Premier Clinical Research /ID# 28168, Spokane, Washington
  - Komorous, Tacoma, WA /ID# 42007, Tacoma, Washington
  - Eastern Washington Dermatology /ID# 17542, Walla Walla, Washington
  - Saoud, Bridgeport, WV /ID# 17135, Bridgeport, West Virginia
  - Mountain State Clinical Research /ID# 28146, Clarksburg, West Virginia
  - Hardy County Medical /ID# 28264, Moorefield, West Virginia
  - Dermatology Assoc of WI /ID# 28142, Appleton, Wisconsin
  - Great Lakes Dermatology /ID# 17061, Pleasant Prairie, Wisconsin
  - Great Lakes Dermatology /ID# 91433, Pleasant Prairie, Wisconsin
  - Aylesworth, Rhinelander, WI /ID# 18322, Rhinelander, Wisconsin
  - Shoreline Skin Specialists, SC /ID# 69771, Sheboygan, Wisconsin
- Austria (11):
  - Duplicate_University Hospital St. Polten /ID# 22842, Sankt Pölten, Lower Austria
  - Medizinische Universitaet Graz /ID# 24263, Graz, Styria
  - Kepler Universitaetsklinikum GmbH /ID# 27922, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH /ID# 17543, Wels, Upper Austria
  - Klinik Landstrasse /ID# 20603, Vienna, Vienna
  - Dr. Harald Maier /ID# 27921, Vienna, Vienna
  - Medizinische Universitaet Wien /ID# 18364, Vienna, Vienna
  - Medizinische Universitaet Wien /ID# 211020, Vienna, Vienna
  - Klinik Hietzing /ID# 17183, Vienna, Vienna
  - Duplicate_Medizinische Universitat Innsbruck,Universitatsklinik fur Innere Mediz /ID# 22844, Innsbruck
  - Landeskrankenhaus Salzburg-Universitätsklinikum der PMU (LKH) /ID# 22843, Salzburg
- Canada (28):
  - Kirk Barber Research, CA /ID# 24204, Calgary, Alberta
  - Stratica Medical /ID# 24266, Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 40199, Surrey, British Columbia
  - Enverus Medical Research /ID# 141448, Surrey, British Columbia
  - University of British Columbia - Eye Care Centre, Vancouver General Hospital /ID# 24223, Vancouver, British Columbia
  - Winnipeg Clinic /ID# 37046, Winnipeg, Manitoba
  - Durondel C.P. Inc. /ID# 28136, Moncton, New Brunswick
  - Karma Clinical Trials /ID# 37049, St. John's, Newfoundland and Labrador
  - Alpha Clinical Research Ctr. /ID# 20581, St. John's, Newfoundland and Labrador
  - Nexus Clinical Research /ID# 79198, St. John's, Newfoundland and Labrador
  - NewLab Clinical Research Inc. /ID# 18360, St. John's, Newfoundland and Labrador
  - Murray, Halifax, CA /ID# 24224, Halifax, Nova Scotia
  - Dermatrials Research /ID# 18363, Hamilton, Ontario
  - The Guenther Dermatology Research Centre /ID# 79196, London, Ontario
  - Lynderm Research Inc. /ID# 18362, Markham, Ontario
  - Entralogix Clinical Research /ID# 79194, Newmarket, Ontario
  - Entralogix Clinical Research /ID# 79197, Newmarket, Ontario
  - Bank on Beauty /ID# 24205, Niagara Falls, Ontario
  - North Bay Dermatology Centre /ID# 28138, North Bay, Ontario
  - SKIN Centre for Dermatology /ID# 79195, Peterborough, Ontario
  - Dr. Jensen Yeung Medicine Professional Corporation /ID# 28141, Toronto, Ontario
  - K. Papp Clinical Research /ID# 28137, Waterloo, Ontario
  - XLR8 Medical Research /ID# 28140, Windsor, Ontario
  - Dr. Isabelle Delorme Inc. /ID# 79193, Drummondville, Quebec
  - Innovaderm Research Inc. /ID# 18866, Montreal, Quebec
  - Centre de Dermatologie Maizerets /ID# 20515, Québec, Quebec
  - Centre de Recherche dermatologique du Quebec Metropolitain /ID# 18361, Québec, Quebec
  - Dr. Beatrice Wang /ID# 18359, Westmount, Quebec
- Czechia (9):
  - Fakultni Nemocnice Brno /ID# 27927, Brno
  - Fakultni nemocnice u sv. Anny v Brne /ID# 37062, Brno
  - Fakultni nemocnice Hradec Kralove /ID# 40201, Hradec Králové
  - Fakultni nemocnice Olomouc /ID# 27930, Olomouc
  - Duplicate_Univ Hosp, Plzen, CZ /ID# 27924, Pilsen
  - Duplicate_Vseobecna fakultni nemoc Praze /ID# 25907, Prague
  - Duplicate_Vseobecna fakultni nemoc Praze /ID# 27933, Prague
  - Vseobecna fakultni nemocnice v Praze /ID# 28269, Prague
  - Krajska zdravotni a.s. Masarykova nemocnice v Usti nad Labem o.z. /ID# 27923, Ústí nad Labem
- Denmark (4):
  - Bispebjerg and Frederiksberg Hospital /ID# 24271, Copenhagen NV, Capital Region
  - Herlev Hospital /ID# 20602, Herlev, Capital Region
  - Aarhus University Hospital /ID# 18357, Aarhus N, Central Jutland
  - Hudklinikken /ID# 20729, Herning
- France (16):
  - Chu de Nice-Hopital L'Archet Ii /Id# 27936, Nice, Alpes-Maritimes
  - HCL - Hopital Lyon Sud /ID# 156129, Pierre-Bénite, Auvergne-Rhône-Alpes
  - HCL - Hopital Lyon Sud /ID# 27940, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU Limoges - Dupuytren 1 /ID# 25904, Limoges, Franche-Comte
  - CHU Bordeaux - Hopital Haut Leveque /ID# 27934, Pessac, Gironde
  - CHRU Lille - Hopital Claude Huriez /ID# 37063, Lille, Hauts-de-France
  - CHU Reims - Hôpital Robert Debre /ID# 37064, Reims, Marne
  - CHU de Nantes, Hotel Dieu -HME /ID# 27944, Nantes, Pays de la Loire Region
  - CHU de SAINT ETIENNE - Hopital Nord /ID# 27942, Saint Priest EN Jarez, Pays de la Loire Region
  - Duplicate_CHU de la miletrie /ID# 25906, Poitiers, Poitou-Charentes
  - CHRU de Besancon - Site Saint-Jacques /ID# 24202, Besançon
  - CHRU Tours - Hopital Trousseau /ID# 28271, Chambray-lès-Tours
  - AP-HM - Hopital Sainte Marguerite /ID# 28270, Marseille
  - Hopital Fournier /ID# 27938, Nancy
  - AP-HP - Hopital Saint-Louis /ID# 24203, Paris
  - Hôpital Charles-Nicolle /ID# 22845, Rouen
- Germany (9):
  - Universitaetsklinik Heidelberg /ID# 20601, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Frankfurt /ID# 19801, Frankfurt am Main, Hesse
  - Universitaetsklinikum Muenster /ID# 37066, Munster, Lower Saxony
  - Universitaetsklinikum Koeln /ID# 27950, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig /ID# 20604, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 22846, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Jena /ID# 19765, Jena, Thuringia
  - Klinikum Ruhr Univ Bochum /ID# 40200, Bochum
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz /ID# 37067, Mainz
- Greece (11):
  - General Hospital Andreas Syggros /ID# 22847, Athens, Attica
  - General Hospital Andreas Syggros /ID# 22848, Athens, Attica
  - General Hospital Andreas Syggros /ID# 25905, Athens, Attica
  - Tzaneio general hospital of Piraeus /ID# 28237, Piraeus, Attica
  - Naval Hospital of Crete /ID# 22849, Crete, Chania
  - University General Hospital of Heraklion PA.G.N.I /ID# 27954, Heraklion, Crete
  - Duplicate_Papageorgiou General Hospital Thessaloniki /ID# 28232, Nea Efkarpia, Thessaloniki
  - Duplicate_Hospital Errikos Ntynan /ID# 28272, Athens
  - General Hospital of Giannitsa /ID# 27951, Giannitsá
  - General Hospital of Katerini /ID# 27953, Katerini
  - Thessaloniki hospital for skin and venereal diseases- Ippokrateio Thessaloniki /ID# 37068, Thessaloniki
- St Vincent's University Hospital /ID# 43149, Elm Park, Dublin, Ireland
- Netherlands (10):
  - Radboud Universitair Medisch Centrum /ID# 24265, Nijmegen, Gelderland
  - Dijklander Ziekenhuis /ID# 18354, Hoorn, North Holland
  - Erasmus Medisch Centrum /ID# 24264, Rotterdam, South Holland
  - Centrum Oosterwal /ID# 18349, Alkmaar
  - ZiekenhuisGroep Twente /ID# 18355, Almelo
  - Academisch Medisch Centrum /ID# 22850, Amsterdam
  - Amphia Ziekenhuis /ID# 20461, Breda
  - Duplicate_Duplicate_Oosterschelde Ziekenhuis /ID# 20462, Goes
  - Spaarne Gasthuis /ID# 22851, Haarlem
  - Diaconessenhuis Voorburg /ID# 18868, Voorburg
- Dr. Reinaldo Rosario Med Offic /ID# 24328, San Juan, Puerto Rico
- Spain (9):
  - Hospital Universitario Germans Trias i Pujol /ID# 17152, Badalona, Barcelona
  - Hospital Duran i Reynals /ID# 18348, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Fundacion Alcorcon /ID# 20723, Alcorcón, Madrid
  - Hospital General Universitario de Alicante Doctor Balmis /ID# 20730, Alicante
  - Hospital Universitari Sagrat Cor - Grupo Quiron Salud /ID# 19767, Barcelona
  - Hospital Clinic de Barcelona /ID# 19803, Barcelona
  - Hospital Universitario de la Princesa /ID# 18867, Madrid
  - Hospital Universitario 12 de Octubre /ID# 18365, Madrid
  - Hospital Clinico Universitario Lozano Blesa /ID# 19763, Zaragoza
- Uppsala University Hospital /ID# 38283, Uppsala, Sweden
- United Kingdom (7):
  - The Royal Free London NHS Foundation Trust /ID# 40205, London, London, City of
  - Guys and St Thomas NHS Foundation Trust /ID# 28273, London, London, City of
  - NHS Greater Glasgow and Clyde /ID# 27956, Glasgow, Scotland
  - Cardiff & Vale University Health Board /ID# 40204, Cardiff, Wales
  - NHS Grampian /ID# 37069, Aberdeen
  - Leeds Teaching Hospitals NHS Trust /ID# 40202, Leeds
  - Northern Care Alliance NHS Group /ID# 40203, Manchester

REFERENCES:
- [Derived] Lynde CW, Alam MS, Ohson K, Gagne-Henley A, Avadisian M, Vender RB. Enhanced Effectiveness of Adalimumab Compared to Topical/Traditional Systemic Agents in the Treatment of Moderate to Severe Plaque Psoriasis: Results from a Canadian Observational Epidemiologic Study (COMPLETE-PS). Dermatol Ther (Heidelb). 2022 Apr;12(4):921-931. doi: 10.1007/s13555-022-00703-3. Epub 2022 Mar 14. PMID 35286612
- [Derived] Menter A, Thaci D, Wu JJ, Abramovits W, Kerdel F, Arikan D, Guo D, Ganguli A, Bereswill M, Camez A, Valdecantos WC. Long-Term Safety and Effectiveness of Adalimumab for Moderate to Severe Psoriasis: Results from 7-Year Interim Analysis of the ESPRIT Registry. Dermatol Ther (Heidelb). 2017 Sep;7(3):365-381. doi: 10.1007/s13555-017-0198-x. Epub 2017 Aug 16. PMID 28815476
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P10-023#additional-resources-section